CLINICAL TRIAL: NCT03620240
Title: An Interactive School Sleep Behavior Modification Program
Brief Title: An Interactive School Sleep Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Michael WL Chee, MBBS, Principle Investigator, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Sleep Education
Record Dates: First submitted 2018-07-24; First posted 2018-08-08 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Education (Experimental): Half of the participants are randomly assigned to the Sleep Education group. These participants will undergo 4 weekly class-based lesson, during which they are educated about sleep.
  Interventions: Behavioral: Sleep Education
- Control (No Intervention): Half of the participants are randomly assigned to the Control group. These participants undergo 4 weekly class-based lessons, during which they are educated about health-related topics, but not about sleep.

INTERVENTIONS:
Behavioral: Sleep Education — Assessing the effectiveness of a Sleep Education Program in improving sleep behaviors in secondary school students.
  Arms: Sleep Education

SUMMARY:
The aim of this study is to improve sleep behavior in secondary school students, through the use of an educational program specifically designed for this purpose. Data will be collected on students' time use, sleep habits, daytime functioning and mood before and after the program to assess if the program is effective in improving students' sleep behavior and corresponding outcomes.

DETAILED DESCRIPTION:
The present study aims to examine the effectiveness of a class-based interactive Sleep Education Program in improving sleep behavior of secondary school students. The Sleep Education Program is designed by sleep experts from our laboratory, and is aimed at educating students about the importance of sleep and good sleep habits, as well as addressing their attitudes towards sleep, in order to encourage behavior change. Participants will be randomly assigned to the Sleep Education Program or a Control Program. All participants will undergo four weekly class-based lessons, which use video presentations, in-class activities, discussions and take-home assignments to deliver the materials. Each lesson has set goals to achieve. Participants in the Sleep Education Program will learn about the importance of sleep, what factors may prevent them from getting enough sleep, how they can manage their time to create more opportunity for sleep, and how they can overcome obstacles to time management. Emphasis will be placed on how sleep affects each student personally, and how each person can benefit from improving sleep. Participants in the Control Program will undergo a similarly structured class-based program, during which they will learn about various general health-related topics. However, the Control Program is designed in such a way that it does not cover any topics related to sleep. Data will be collected from participants from both groups. The following variables are measured: sleep habits, sleep knowledge, daytime functioning, mood and app-tracked time use. Data on all measurements will be collected at three time points: pre-program, immediately post-program and during a 1-month follow-up. Results will be compared between the three time points, as well as between the two groups (Sleep Education Program and Control Program). By comparing results from the Sleep Education Program to the Control Program, we can evaluate the effect of educating students about sleep on improving sleep behavior.

ELIGIBILITY:
Inclusion Criteria:

* Secondary school students
* Currently in year 2

Exclusion Criteria:

* Secondary school students form years other than year 2

Ages: 13 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 205 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Change in actigraphically measured sleep behavior between time 1 (pre-program), time 2 (immediately post-program) and time 3 (at 1-month follow-up), measured for one week in each of the three phases. | 3 times (pre-program, immediately post-program and at 1-month follow-up)
  Bedtime, wake up time, time in bed, total sleep time, sleep efficiency, timing and duration of daytime naps
Change in sleep dairy reported sleep behavior between time 1 (pre-program), time 2 (immediately post-program) and time 3 (at 1-month follow-up), recorded for one week in each of the three phases. | 3 times (pre-program, immediately post-program and at 1-month follow-up)
  Bedtime, wake up time, total sleep time, sleep efficiency, number and duration of nighttime awakenings, number and duration of daytime naps
Change in the level of subjective mood between time 1 (pre-program), time 2 (immediately post-program) and time 3 (at 1-month follow-up), measured once daily with a Mood Rating Scale over the period of one week. | 3 times (pre-program, immediately post-program and at 1-month follow-up)
  Score on the Mood Rating Scale. Range: 1 (extremely bad) to 9 (extremely good). Higher values represent a better outcome.
Change in the level of subjective sleepiness between time 1 (pre-program), time 2 (immediately post-program) and time 3 (at 1-month follow-up), measured once daily with the Karolinska Sleepiness Scale over the period of one week. | 3 times (pre-program, immediately post-program and at 1-month follow-up)
  Score on the Karolinska Sleepiness Scale. Range: 1 (extremely alert) to 9 (extremely sleep, fighting sleep). Lower values represent a better outcome.
Change in sleep knowledge between time 1 (pre-program), time 2 (immediately post-program) and time 3 (at 1-month follow-up), measured with a sleep knowledge questionnaire. | 3 times (pre-program, immediately post-program and at 1-month follow-up)
  Score on the sleep knowledge questionnaire. Range: 0 (all incorrect answers) to 12 (all correct answers). Higher values represent a better outcome.
Change in time use between time 1 (pre-program), time 2 (immediately post-program) and time 3 (at 1-month follow-up), measured daily with a time use diary over the period of one week. | 3 times (pre-program, immediately post-program and at 1-month follow-up)
  Amount of time spent on each activity
Relationship between sleep and time use. | 3 times (pre-program, immediately post-program and at 1-month follow-up)
  Amount of time spent on each activity, measured with a time use diary, correlated with sleep variables, measured with actigraphy and a sleep diary.

CONTACTS AND LOCATIONS:
Overall Officials: Michael WL Chee, MBBS, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Duke-NUS Medical School, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Rijn E, Koh SYJ, Ng ASC, Vinogradova K, Chee NIYN, Lee SM, Lo JC, Gooley JJ, Chee MWL. Evaluation of an interactive school-based sleep education program: a cluster-randomized controlled trial. Sleep Health. 2020 Apr;6(2):137-144. doi: 10.1016/j.sleh.2019.10.006. Epub 2019 Dec 4. PMID 31812609

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT03620240/Prot_SAP_000.pdf